CLINICAL TRIAL: NCT04450953
Title: A Randomized Crossover Clinical Trial Regarding the Blockage of the Mineralocorticoid Receptor Using Eplerenone on the Evolution of Arterial Stiffness in Kidney Patients One Year After Transplant
Brief Title: The Effect of Eplerenone on the Evolution of Vasculopathy in Renal Transplant Patients.
Acronym: EVATRAN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr. Nicolas GIRERD, Study Chair, Central Hospital, Nancy, France
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019-004243-74
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Kidney Transplantation for More Than One Year; Patients with a Kidney Transplantation on Cyclosporine
MeSH Terms: interventions — Eplerenone; Cross-Over Studies

STUDY DESIGN:
Intervention Model Description: * Arm A in which they will receive eplerenone 50mg/day taken orally for 6 months, followed by a 8 to 10 weeks wash-out period, then a 6-month period without eplerenone, until the end of the study.
  * arm B where they will be eplerenone-free for 6 months, followed by a 8 to 10 weeks wash-out period, then a 6-month period in which they will receive eplerenone 50 mg/day as a single dose taken orally.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eplerenone group A (cross over design) (Active Comparator): Patient will receive eplerenone 50mg/day taken orally for 6 months, followed by a 8 to 10 weeks wash-out period, then a 6-month period without eplerenone, until the end of the study.
  Interventions: Drug: Eplerenone 50mg/day (cross over design); Other: Period without eplerenone (cross over design)
- Eplerenone group B (cross over design) (Active Comparator): Eplerenone-free for 6 months, followed by a 8 to 10 weeks wash-out period, then a 6-month period in which patients will receive eplerenone 50 mg/day as a single dose taken orally.
  Interventions: Drug: Eplerenone 50mg/day (cross over design); Other: Period without eplerenone (cross over design)

INTERVENTIONS:
Drug: Eplerenone 50mg/day (cross over design) — Eplerenone 50mg/day for 6 months followed
Other: Period without eplerenone (cross over design) — 6-month period without eplerenone

SUMMARY:
Cardiovascular (CV) pathologies are the leading cause of death in kidney transplant patients.Arterial stiffness is a prognostic factor for CV mortality in kidney transplantation. Despite a reduced CV risk in transplant kidney patients in comparison to patients in dialysis, CV mortality among kidney transplant patients is much higher than the general population.

After renal transplantation, the cardiac and vascular anomalies observed in chronic end-stage renal disease are partially improved because of restored normal kidney function and withdrawal from dialysis.

However, patients are exposed to immunosuppressive drugs, in particular calcineurin inhibitors, which can be associated with vascular toxicity, either directly or by promoting the appearance of hypertension, diabetes, or dyslipidemia.The pathophysiology of arterial stiffness in kidney transplantation is complex and multifactorial.

Calcineurin inhibitors are likely to play an important role in the persistence of increased arterial stiffness in transplant patients in whom renal function has been restored. Indeed, the discontinuation of anti-calcineurins in favour of other molecules .is associated with a decrease of arterial stiffness.

Preclinical work has shown that the vascular toxicity of cyclosporine is mediated by activation of the mineralocorticoid receptor in smooth muscle cells. The involvement of the mineralocorticoid receptor in the onset of arterial stiffness is also well demonstrated in non-transplanted subjects.

Blocking the mineralocorticoid receptor in patients under cyclosporine may reduce their arterial stiffness and in and consequently improve their CV prognosis.

Studies have show a good safety in kidney transplant patients. This pilot study proposes to examine, for the first time, the impact of treatment with a mineralocorticoid receptor antagonist on the evolution of arterial stiffness in renal transplant patients on calcineurin inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 50 years of age;
* Patient who had a kidney transplant at least one year prior to inclusion;
* Patient on cyclosporine;
* Patient whose clinical-biological state has been stable for at least 3 months: no change in treatment with an impact on blood pressure (excluding immunosuppressive drug) for 3 months, no acute rejection diagnosed within 3 months;
* Patient with a glomerular filtration rate estimated according to the formula CKD-EPI ≥30mL/min/1.73m2;
* Patient with a peripheral PAS≥110mmHg, irrespective of the presence or not of an antihypertensive therapy (including ACE inhibitors or sartan) ;
* Patient with signed informed consent;
* Patient affiliated with or beneficiary of a social security system.

Exclusion Criteria:

* Patient with documented kalemia ≥ 5mmol/L in the last 15 days;
* Patient undergoing mineralocorticoid receptor antagonism or with a formal indication to receive this treatment;
* Bicarbonate blood level <20mmol/L with or without documented supplementation in the last 15 days.
* Indication for a combination of ACE inhibitor and sartan (each of which is authorized separately);
* Patient under another potassium sparing diuretics;
* Patient under digoxine;
* Sodium polystyrene sulfonate contraindication;
* Known hypersensitivity or allergy to eplerenone and its excipients;
* Patient with severe hepatic impairment (Child-Pugh Class C);
* Patient under CYP3A4 inhibitor;
* know intolerance to Galactose, a Lapp lactase deficiency or galactose malabsorption syndrome;
* Patient participating in other interventional research;
* Woman with a desire of pregnancy within 15 months;
* Woman of childbearing age without effective contraception;
* Persons referred to in Articles L. 1121-5, L. 1121-7 and L1121-8 of the Public Health Code :
* Pregnant women, parturient women or nursing mothers ;
* Adult person subject to a legal protection measure (guardianship, curator, judicial safeguard);
* Adults person who is unable to give consent and who is not subject to a legal protection measure;
* Persons deprived of their liberty by a judicial or administrative decision;
* Persons subject to psychiatric care pursuant to articles L. 3212-1 and L. 3213-1.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Evolution of pulse wave velocity (PWV in m/s) adjusted to the blood pressure | After 6 months of treatment with eplerenone

SECONDARY OUTCOMES:
Evolution of Central Systolic Blood Pressure (CSPc) | After 6 months of treatment with eplerenone
Evolution of central Diastolic Blood Pressure (CDAb) | After 6 months of treatment with eplerenone
Evolution of Central Pulsed Pressure (CPp) | After 6 months of treatment with eplerenone
Evolution of Augmentation index (Aix in %) | After 6 months of treatment with eplerenone
Evolution peripheral systolic blood pressure (PASp in mmHg) | After 6 months of treatment with eplerenone
Evolution of peripheral diastolic blood pressure (PADp in mmHg) | After 6 months of treatment with eplerenone
Evolution of peripheral pulse pressure (PPp in mmHg) | After 6 months of treatment with eplerenone
Evolution of Intima-media thickness (in mm) | After 6 months of treatment with eplerenone
Evolution of left ventricular mass (LVM in g/m2) | After 6 months of treatment with eplerenone
Evolution of biological markers of oxidative stress (plasma Isoprostane) | After 6 months of treatment with eplerenone
Evolution of biological markers of oxidative stress (Malondialdehyde) | After 6 months of treatment with eplerenone
Evolution of Biological markers of endothelial dysfunction (endothelin) | After 6 months of treatment with eplerenone
Evolution of biological markers of endothelial dysfunction (soluble endothelium selectin (sE-selectin)) | After 6 months of treatment with eplerenone
Evolution of biological markers of endothelial dysfunction (von Willebrand factor) | After 6 months of treatment with eplerenone
Evolution of graft function | After 6 months of treatment with eplerenone
  measured by creatinine (in micromol/L) with estimation of glomerular filtration rate (eGFR in mL/min/1.73m2 ) according to the CKD-EPI formula.
Evolution of proteinuria | After 6 months of treatment with eplerenone
  measured by the ratio proteinuria/creatinuria (in mg/g)
Percentage of patients with DFG ≥ 90, 60-89, 45-59, 30-44, 15-29 <15ml/min/1,73m2 | After 6 months of treatment with eplerenone
Percentage of patient with ratio proteinuria/creatinuria (en mg/g) <500 ; 500-1000, 1000-2000, 2000-3000, >3000 | After 6 months of treatment with eplerenone
hyperkalemia occurence ≥ 5.5 mmol/L | during 6 month of treatment with eplerenone
Number of hyperkalemia | during 6 month of treatment with eplerenone
  number of hyperkalemias during hyperkalemia follow-up between 5 - 5.49; 5.5 - 6; >6mmol/L
increase of creatinine of more than 50% | during 6 month of treatment with eplerenone
  Evaluation of risk of acute renal failure defined as an increase in creatinine of more than 50%

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GIRERD, MD-Phd, Study Chair — Central Hospital, Nancy, France; Sophie GIRERD, MD-PhD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Derived] Simon A, Girerd N, Jaisser F, Bozec E, Lepage X, Merckle L, Rossignol P, Frimat L, Girerd S. EVATRAN (The Effect of Eplerenone on the Evolution of Vasculopathy in Renal Transplant Patients): study protocol for a cross-over randomized controlled trial. Trials. 2025 Nov 7;26(1):479. doi: 10.1186/s13063-025-09187-w. PMID 41204172
- [Derived] Natale P, Mooi PK, Palmer SC, Cross NB, Cooper TE, Webster AC, Masson P, Craig JC, Strippoli GF. Antihypertensive treatment for kidney transplant recipients. Cochrane Database Syst Rev. 2024 Jul 31;7(7):CD003598. doi: 10.1002/14651858.CD003598.pub3. PMID 39082471